CLINICAL TRIAL: NCT00855400
Title: Phase I/II Clinical Trial on the Use of Autologous Bone Marrow Stem Cells in Amyotrophic Lateral Sclerosis
Brief Title: Clinical Trial on the Use of Autologous Bone Marrow Stem Cells in Amyotrophic Lateral Sclerosis
Acronym: CMN/ELA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Collaborators: Carlos III Health Institute (Other Government); Hospital Universitario Virgen de la Arrixaca (Other); Hospital General Universitario Morales Meseguer (Other); Diógenes Foundation (Other)
Responsible Party: Javier Júdez Gutiérrez, Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMN/ELA; EudraCT number: 2006-003096-12; ISCIII: EC07/90762
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Bone marrow; Stem cells; Autologous; Safety
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Laminectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transplant (Experimental): T3-T4 laminectomy and bone marrow ficoll separated mononuclear autologous cells intraspinal transplantation
  Interventions: Procedure: Laminectomy and bone marrow stem cells transplantation; Procedure: Autologous bone marrow cells collection

INTERVENTIONS:
Procedure: Laminectomy and bone marrow stem cells transplantation — T3-T4 laminectomy and bone marrow ficoll separated mononuclear autologous cells intraspinal transplantation
Procedure: Autologous bone marrow cells collection — Autologous bone marrow cells collection under sedation. Sixty mL are obtained and processed through a ficoll gradient.

SUMMARY:
The purpose of this clinical trial is to asses the feasibility and the security of the intraspinal infusion of autologous bone marrow stem cells for the treatment of Amyotrophic Lateral Sclerosis patients.

DETAILED DESCRIPTION:
Patients with Amyotrophic Lateral Sclerosis (ALS) typically endure a progressive paralysis due to the continued loss of motoneurons that leads them to death in less than 5 years. No treatment has changed its natural history. Intraspinal injections of bone marrow mononuclear cells (MNC) have been able to ameliorate the course of ALS in murine models, acting as pumps of trophic factors that keep the motoneurons functional. We have designed a phase I/II clinical trial to check the feasibility of this approach in humans.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose established following the World Federation of Neurology criteria
* More than 6 and less than 36 months of evolution of the disease
* Medullar onset of the disease
* More than 20 and less than 65 years old
* Forced Vital Capacity equal or superior to 50%
* Total time of oxygen saturation <90% inferior to 2% of the sleeping time
* Signed informed consent

Exclusion Criteria:

* Neurological or psychiatric concomitant disease
* Need of parenteral or enteral nutrition through percutaneous endoscopic gastrostomy or nasogastric tube
* Concomitant systemic disease
* Treatment with corticosteroids, immunoglobulins or immunosuppressors during the last 12 months
* Inclusion in other clinical trials
* Unability to understand the informed consent

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-02; Primary Completion 2009-10 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity | Every 3 months

SECONDARY OUTCOMES:
ALS-FRS, MRC and Norris scales | Every 3 months
Absence of adverse events | Every week / month depending on the study phase

CONTACTS AND LOCATIONS:
Overall Officials: Jose Maria Moraleda Jiménez, M.D. Ph.D., Study Director — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia, Spain

REFERENCES:
- [Derived] Blanquer M, Moraleda JM, Iniesta F, Gomez-Espuch J, Meca-Lallana J, Villaverde R, Perez-Espejo MA, Ruiz-Lopez FJ, Garcia Santos JM, Bleda P, Izura V, Saez M, De Mingo P, Vivancos L, Carles R, Jimenez J, Hernandez J, Guardiola J, Del Rio ST, Antunez C, De la Rosa P, Majado MJ, Sanchez-Salinas A, Lopez J, Martinez-Lage JF, Martinez S. Neurotrophic bone marrow cellular nests prevent spinal motoneuron degeneration in amyotrophic lateral sclerosis patients: a pilot safety study. Stem Cells. 2012 Jun;30(6):1277-85. doi: 10.1002/stem.1080. PMID 22415951